CLINICAL TRIAL: NCT00164346
Title: Neurocognitive Habilitation for Children With FAS/ARND
Brief Title: Neurocognitive Habilitation for Children With Fetal Alcohol Syndrome (FAS)/Alcohol-Related Neurodevelopmental Disorder (ARND)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Children's Research Triangle (Unknown)
Responsible Party: Jacquelyn Bertrand, CDC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CDC-NCBDDD-3710; U84/CCU520164-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Fetal Alcohol Syndrome; Alcohol-related Neurodevelopmental Disorder
Keywords: fetal alcohol syndrome (FAS); alcohol-related neurodevelopmental disorder (ARND)
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

INTERVENTIONS:
Behavioral: neurocognitive habilitation

SUMMARY:
Children will receive comprehensive evaluations through the Children's Research Triangle (CRT) clinical program. The assessment for the child will be in accordance with the protocol developed by Astley and Clarren as performed by one of the clinic pediatricians and final diagnosis will be according to Institute of Medicine (IOM) criteria. Children will be randomized into either a Treatment or Control group. The Treatment group will receive (in addition to standard referrals) neurocognitive habilitation and psychotherapy services as well as parent psychoeducation. The Control group will be referred for intervention through existing community and school-based agencies.

DETAILED DESCRIPTION:
Neurocognitive habilitation, based on the traumatic brain injury literature for teaching compensatory skills, will be the primary intervention. Interventions will be individually designed and delivered through individual therapy sessions. Audiotapes will augment the sessions to facilitate implementation of strategies in the home environment. Didactic therapy will be used to foster appropriate interactions and relationships between parent and child. Children will participate in 8-week group sessions that will include neurocognitive exercises, homework sessions, and possibly group psychotherapy. An educational specialist will provide school and legal advocacy services as well as observations of the child in the classroom that could lead to educational modifications.

Parent Component: Family education programs and parent support groups using psychoeducational approaches will be the means of intervening with parent behaviors. Parents will be instructed on becoming advocates for their child. Groups of 8 to 12 parents will meet for one 2-hour session per week for 8 weeks. Each session will include:

1. neurocognitive exercises (relaxation);
2. specific topic discussions; and
3. general support.

During the last hour of the final two weeks of the program, parent and children will be combined to practice learned techniques. Children and parents will participate in monthly "booster" sessions.

Evaluation Plan: Treatment and control groups will be compared using pre- and post-test measures. Post-tests will be at the conclusion of the intervention, as well as at 12, and 24-month follow-ups. Process and outcome measures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years
* Children in the care of Illinois foster care

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2002-01; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
foster care placement stability

CONTACTS AND LOCATIONS:
Overall Officials: Ira Chasnoff, MD, Principal Investigator — Children's Research Triangle
Locations (1):
- Children's Research Triangle, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wells AM, Chasnoff IJ, Schmidt CA, Telford E, Schwartz LD. Neurocognitive habilitation therapy for children with fetal alcohol spectrum disorders: an adaptation of the Alert Program(R). Am J Occup Ther. 2012 Jan-Feb;66(1):24-34. doi: 10.5014/ajot.2012.002691. PMID 22251828
- [Derived] Chasnoff IJ, Wells AM, Telford E, Schmidt C, Messer G. Neurodevelopmental functioning in children with FAS, pFAS, and ARND. J Dev Behav Pediatr. 2010 Apr;31(3):192-201. doi: 10.1097/DBP.0b013e3181d5a4e2. PMID 20375733